CLINICAL TRIAL: NCT01061996
Title: An Open Label Evaluation of the Safety and Efficacy of Basiliximab Maintenance in Ulcerative Colitis
Brief Title: Basiliximab Maintenance in Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Cerimon Pharmaceuticals (Industry)
Responsible Party: Shaily J. Reichert, Cerimon Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSX-002
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Basiliximab — Study Drug: basiliximab 40 mg, given as a short intravenous infusion Dosing Schedule: once every 4 weeks Concomitant Therapy: Oral corticosteroids (prednisone or equivalent) will be tapered during the first few months of the study participation Duration of Study Participation: The duration of individual study participation will vary.
  Other Names: Simulect

SUMMARY:
Primary Objective Safety: assess the safety of basiliximab 40 mg, given every 4 weeks, in subjects with ulcerative colitis who completed previous basiliximab studies.

Secondary Objectives: evaluate the efficacy and assess the immunogenicity of this multiple-dose maintenance regimen in this population

ELIGIBILITY:
Inclusion Criteria:

1. Previously met eligibility criteria in the previous basiliximab UC study
2. Must have a total Mayo score at entry consistent with clinical response or clinical remission.
3. Signed a current IRB/IEC-approved informed consent form
4. Females of childbearing potential must use an effective birth control method, and be willing to continue birth control during the study, and for 4 months after the last dose of study drug.
5. Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months before study entry, hysterectomy, or bilateral oophorectomy at least 2 months before study entry) or post-menopausal for at least 2 years.

Exclusion Criteria:

1. Subject is severely ill, as evidenced by more than 6 episodes of loose stools, all of them bloody, during a 24-hour period within the prior 7 days, concurrent with any of the following systemic features:

   * Heart rate > 90 beats/min at rest
   * Temperature > 37.8 degrees C
   * Hemoglobin < 10.5 g/dL
2. Subject is currently receiving a restricted/prohibited concomitant medication
3. Subject has undergone colectomy (total, or subtotal)
4. Subject is pregnant or breast-feeding
5. Prior noncompliance with previous study visit schedule and requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess the safety of basiliximab in subjects with ulcerative colitis | 1 year

SECONDARY OUTCOMES:
Evaluate the efficacy and assess the immunogenicity of t his multiple-dose maintenance regimen in this population | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shaily J. Reichert, Study Director — Cerimon Pharmaceuticals
Locations (1):
- Bristol, United Kingdom